CLINICAL TRIAL: NCT05997732
Title: Sympathetic Neurovascular Transduction: Role of Adrenergic Receptors and Sex Differences
Acronym: STARS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00126600
Record Dates: First submitted 2023-08-02; First posted 2023-08-18 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Vasoconstriction; Vasodilation
Keywords: sympathetic nerve activity; sex differences; adrenergic receptors; neurovascular transduction
MeSH Terms: conditions — Aneurysm | interventions — Phenylephrine; Isoproterenol; Norepinephrine; Propranolol; Phentolamine

STUDY DESIGN:
Intervention Model Description: Participants will complete three pharmacological conditions, and serve as their own controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Condition (Experimental): Normal saline will be infused through the brachial artery catheter at the same calculated rate as propranolol + phentolamine in the α+β-blockade condition to control for volumetric effects.
  Interventions: Drug: Phenylephrine Hydrochloride; Drug: Isoproterenol Hydrochloride; Drug: Norepinephrine Bitartrate
- β-Adrenergic Blockade (Experimental): β-adrenoreceptors will be blocked locally in the forearm using propranolol. Normal saline will be co-infused at the calculated rate of phentolamine in the α+β-blockade condition to control for volumetric effects.
  Interventions: Drug: Norepinephrine Bitartrate; Drug: Propranolol Hydrochloride
- α+β-Adrenergic Blockade (Experimental): α-adrenoreceptors will be blocked locally in the forearm using phentolamine. Propranolol will be co-infused to maintain β-blockade.
  Interventions: Drug: Phentolamine Mesylate; Drug: Phenylephrine Hydrochloride; Drug: Isoproterenol Hydrochloride; Drug: Propranolol Hydrochloride

INTERVENTIONS:
Drug: Phenylephrine Hydrochloride — Participants will receive three incremental doses via the brachial artery catheter to assess α1-adrenoreceptor mediated vasoconstriction.
  Arms: Control Condition
Drug: Isoproterenol Hydrochloride — Participants will receive four incremental doses via the brachial artery catheter to assess β-adrenoreceptor mediated vasodilation.
  Arms: Control Condition
Drug: Norepinephrine Bitartrate — Participants will receive three incremental doses via the brachial artery catheter to assess nonspecific adrenoreceptor activation.
  Arms: Control Condition; β-Adrenergic Blockade
Drug: Propranolol Hydrochloride — Propranolol will be continuously infused through the brachial artery catheter to induce β-adrenergic blockade locally in the forearm.
  Arms: β-Adrenergic Blockade
Drug: Phentolamine Mesylate — Phentolamine will be continuously infused through the brachial artery catheter to induce α-adrenergic blockade locally in the forearm.
  Arms: α+β-Adrenergic Blockade
Drug: Phenylephrine Hydrochloride — Participants will receive one dose via the brachial artery catheter to evaluate the effectiveness of the α-adrenergic blockade.
  Arms: α+β-Adrenergic Blockade
Drug: Isoproterenol Hydrochloride — Participants will receive one dose via the brachial artery catheter to evaluate the effectiveness of the β-adrenergic blockade.
  Arms: α+β-Adrenergic Blockade
Drug: Propranolol Hydrochloride — Propranolol will be continuously co-infused with phentolamine to maintain the β-adrenergic blockade.
  Arms: α+β-Adrenergic Blockade

SUMMARY:
The main purpose of this interventional study is to examine differences in resting blood pressure control between healthy males and females. The main questions it aims to answer are:

1. Are there sex differences in the communication between the sympathetic nervous system (also known as the "fight or flight" response) and peripheral blood vessels (which influence systemic blood pressure)?
2. What is the role of specific vascular receptors that respond to sympathetic signals, and is it different between males and females?

Participants will complete one study visit of approximately 3 hours where they will:

* Have a blood sample taken to measure circulating sex hormone and sympathetic transmitters.
* Receive very small doses of medications commonly used to adjust blood pressure through an artery in their arm. The effects of these medications will be short-acting and localized to the forearm.
* Have their sympathetic nervous activity directly measured through two very small needles (similar to acupuncture needles) in the side of their leg.
* Have their blood pressure and heart rate recorded, and forearm blood flow measured using ultrasound.

DETAILED DESCRIPTION:
Blood pressure is in part regulated by activity of your sympathetic nervous system (also known as your "fight or flight" response). Sympathetic nerve activity affects the size of your blood vessels, which in turn will affect your blood pressure. This communication between sympathetic impulses and the resulting change in vascular resistance is termed "sympathetic neurovascular transduction". In other words, transduction represents the reactivity of the blood vessels in response to individual sympathetic bursts of activity.

Males and females regulate their blood pressure in different ways; for example, females tend to have lower blood pressure and sympathetic nerve activity than males. Females also appear to have less constriction of their blood vessels in response to stress. This may be due to differences in the receptors which are activated by the sympathetic nervous system. These receptors are called α and β-adrenergic receptors and are located on vascular smooth muscle cells. They respond to sympathetic neurotransmitters such as norepinephrine in opposite directions: α-adrenoreceptors cause vasoconstriction (and an increase in vascular resistance), and β-adrenoreceptors cause vasodilation (and a decrease in vascular resistance) in part through the endothelium-dependent nitric oxide pathway.

Current evidence suggests that β-adrenergic receptors are more sensitive in females and contribute to paradoxical vasodilation when α-adrenergic receptors are stimulated by norepinephrine from sympathetic bursts. It has also been suggested that estrogen interacts with adrenergic receptors, contributing to this sex difference. This study will contribute to the understanding of sex differences in cardiovascular physiology and may have implications for clinical cardiovascular conditions.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 18-40 years
* No diagnosed medical history of cardiovascular, respiratory, nervous system, or metabolic disease.
* Females must be pre-menopausal.
* Prior to study visit: abstained from caffeine, alcohol, strenuous exercise, and medication not taken regularly for at least 12 hours.

Exclusion Criteria:

* Current diagnosis of cardiovascular, respiratory, nervous system, or metabolic disease that may impact blood pressure regulation. This will be assessed on a case-by-case basis by the study physician.
* Participants with bleeding or clotting disorders, or those currently taking blood thinners.
* Participants currently taking beta-agonist inhalers i.e. Ventolin (at least not in the last 24 hours).
* Females who are pregnant, confirmed by a pregnancy test.
* Females who have are less than 1 year postpartum or are breastfeeding.
* Females who are post-menopausal.
* Participants that are classified as obese (body mass index > 30 kg ⋅ m2).
* Have a history of smoking regularly in the last 6 months (but nicotine substitutes (i.e. patch, gum) are not an exclusion criteria).
* Those with a known allergy to sulfites, or other components of the supplied solution of study drugs.
* Participants taking medications that are contraindicated with any of the study drugs, such as monoamine oxidase (MAO) inhibitors or tricyclic antidepressants.
* Participants who have not adhered to the pre-testing guidelines related to diet, alcohol or exercise will not be excluded, but will be rescheduled for a different day. This is to reduce experimental variability.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Forearm blood flow | 10 minutes per condition + 2 minutes per agonist dose = 60 minutes
  Measured during resting baseline; changes during phenylephrine, isoproterenol, and norepinephrine infusion to determine agonist sensitivity.
Forearm vascular resistance | 10 minutes per condition + 2 minutes per agonist dose = 60 minutes
  Measured during resting baseline; changes during phenylephrine, isoproterenol, and norepinephrine infusion to determine agonist sensitivity.
Forearm vascular conductance | 10 minutes per condition + 2 minutes per agonist dose = 60 minutes
  Measured during resting baseline; changes during phenylephrine, isoproterenol, and norepinephrine infusion to determine agonist sensitivity.
Arterial blood pressure | 10 minutes per condition + 2 minutes per agonist dose = 60 minutes
  Measured during resting baseline; changes during phenylephrine, isoproterenol, and norepinephrine infusion to determine agonist sensitivity.
Muscle sympathetic nerve activity | 10 minutes per condition = 30 minutes
  Resting baseline
Circulating sex hormone concentrations | 2 minutes
  Blood samples
Circulating sympathetic neurotransmitter concentrations | 2 minutes
  Blood sample

SECONDARY OUTCOMES:
Arterial-venous blood gas concentrations | 2 minutes per sample = 6 minutes
  Blood sample during each condition

CONTACTS AND LOCATIONS:
Overall Officials: Sean van Diepen, MD, MSc, Principal Investigator — University of Alberta; Craig Steinback, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Hart EC, Charkoudian N, Wallin BG, Curry TB, Eisenach JH, Joyner MJ. Sex differences in sympathetic neural-hemodynamic balance: implications for human blood pressure regulation. Hypertension. 2009 Mar;53(3):571-6. doi: 10.1161/HYPERTENSIONAHA.108.126391. Epub 2009 Jan 26. PMID 19171792
- [Background] Steinback CD, Fraser GM, Usselman CW, Reyes LM, Julian CG, Stickland MK, Chari RS, Khurana R, Davidge ST, Davenport MH. Blunted sympathetic neurovascular transduction during normotensive pregnancy. J Physiol. 2019 Jul;597(14):3687-3696. doi: 10.1113/JP277714. Epub 2019 Jun 13. PMID 31106429
- [Background] Fairfax ST, Holwerda SW, Credeur DP, Zuidema MY, Medley JH, Dyke PC 2nd, Wray DW, Davis MJ, Fadel PJ. The role of alpha-adrenergic receptors in mediating beat-by-beat sympathetic vascular transduction in the forearm of resting man. J Physiol. 2013 Jul 15;591(14):3637-49. doi: 10.1113/jphysiol.2013.250894. Epub 2013 May 7. PMID 23652594
- [Background] Dinenno FA, Eisenach JH, Dietz NM, Joyner MJ. Post-junctional alpha-adrenoceptors and basal limb vascular tone in healthy men. J Physiol. 2002 May 1;540(Pt 3):1103-10. doi: 10.1113/jphysiol.2001.015297. PMID 11986395
- [Background] Hissen SL, Taylor CE. Sex differences in vascular transduction of sympathetic nerve activity. Clin Auton Res. 2020 Oct;30(5):381-392. doi: 10.1007/s10286-020-00722-0. Epub 2020 Aug 31. PMID 32865664